CLINICAL TRIAL: NCT05319405
Title: A Pilot Investigation of the Effectiveness of the Sana Device in Management of PTSD: A Blinded Randomized Controlled Trial
Brief Title: Effectiveness of Sana Treatment in Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Health (Industry)
Collaborators: Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00119759; CLN-013-A (Other: Sana Health, Inc.)
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-11

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Parallel 2-arm study in which participants will be randomly assigned to either Sana plus Treatment as Usual (Sana+TAU) or Treatment as Usual (TAU)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sana plus Treatment as Usual (Active Comparator): Subjects will be loaned a Sana Device to use for 28 days and will also receive mental health care through the Ralph H. Johnson VA Medical Center.
  Interventions: Device: Sana Device
- Treatment as Usual (No Intervention): Subjects will receive mental health care at the Ralph H. Johnson VA Medical Center or community-based outpatient clinic (CBOC).

INTERVENTIONS:
Device: Sana Device — Externally worn mask that physically contacts the skin of the face. The Sana Device delivers Audio Visual Stimulation (AVS) in the form of coordinated pulses of light (through closed eyelids) and sound at various frequencies.
  Arms: Sana plus Treatment as Usual

SUMMARY:
The purpose of this study is to assess the effectiveness of the Sana Device when added to Treatment as Usual in participants with a diagnosis of post-traumatic stress disorder (PTSD)

DETAILED DESCRIPTION:
This is a study designed to assess the effectiveness of the Sana Device when added to Treatment as Usual in participants with a diagnosis of post-traumatic stress disorder (PTSD) on severity of symptoms as measured by CAPS-5. We will use a 2-arm repeated measures randomized controlled design in which participants will be randomly assigned to either Sana plus Treatment as Usual (Sana+TAU) or Treatment as Usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Having served, or are currently serving, in the US military with a VA CPRS record.
* Willing to and capable of providing written electronic informed consent prior to the conduct of any study-related procedures.
* Adults, of any sex or gender, 18 to 65 years of age.
* Diagnosis of PTSD as determined by a Clinician Administered PTSD Scale for DSM-5 (CAPS-5) clinical interview or CAPS-5 severity ≥ 25.
* Must be in good physical health based on self-report.
* Any psychotropic drug therapy regimen must be stable (unchanging) for at least 4 weeks prior to enrollment and remain steady throughout the study.
* Willing and able to comply with the study requirements, complete study assessments, and participate at scheduled times for the duration of the study.
* Able to understand, speak, and read English sufficient for the completion of study assessments.
* Provision of appropriate storage and charging for study equipment in a generally safe and dry condition.

Exclusion Criteria:

* Pregnant, intending to become pregnant, or lactating females as self-reported.
* History or presence of photo-sensitive epilepsy or other photo-sensitive conditions as self-reported.
* History or presence of condition(s) that may affect balance, such as seizure disorders or vertigo as self-reported.
* History or presence of severe and continuous tinnitus, at investigator discretion
* Surgery or trauma requiring rehabilitation within the last 12 weeks as self-reported. Presence of cancer pain, acute pain following injury or other severe pain that would be anticipated to change during the course of the study, at discretion of the investigator.
* Vision impairments that affect perception of light, color, or brightness in one or both eyes, and differences in visual perception between eyes, per patient self-report.
* Deafness in one or both ears, perceived differences in hearing between ears, per patient self-report.
* Current ear or eye infection, untreated allergies, or acute illness that may affect eyes or hearing (e.g., due to congestion), per patient self-report.
* Presence of inflammation or broken skin around the eyes in the area of the mask, per patient self-report.
* Presence of narcolepsy or untreated sleep apnea, per patient self-report. Note: presence of sleep apnea is permitted, so long as patients feel comfortable to use both apnea mask and Sana device in conjunction.
* Participation in any other clinical study in which medication(s) are being delivered or have used an investigational drug or device within the last 30 days.
* Any pending legal action that could prohibit participation or compliance in the study, per patient self-report.
* Recent history of or current evidence of suicidal intent or active suicidal behavior based on patient self-report at investigator discretion.
* Significant medical conditions or other circumstances which, in the opinion of the investigator, would preclude compliance with the protocol, adequate cooperation in the study or obtaining informed consent, or may prevent the patient from safely participating in study.
* Employment by the investigator or the study site, with direct involvement in the proposed study or other studies under the direction of the investigator or study site, or a family member of an employee or of the investigator.
* Use of drugs that can produce hallucinogenic effects (i.e., Ketamine or psilocybin mushrooms) within the past 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
To examine the difference between Sana plus Treatment as Usual (Sana+TAU) and Treatment as Usual (TAU) on changes in PTSD symptoms as measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5) after 28 days. | Baseline and Day 28
  A 30-item structured interview that can be used to diagnosis and assess PTSD symptoms and severity.

SECONDARY OUTCOMES:
To examine the difference between Sana+TAU and TAU on changes in PTSD symptoms as measured by the PTSD Checklist - 20-item scale for DSM-5 (PCL-5) after 28 days. | Baseline, Days 14 and 28
  A 20-item self-reported measure that assesses the 20 DSM-5 symptoms of PTSD.
To examine the difference between Sana+TAU and TAU on anxiety symptoms as measured by the Generalized Anxiety Disorder 7-item scale (GAD-7) after 28 days. | Baseline, Days 14 and 28
  The GAD-7 is a self-reported questionnaire for screening and measuring severity of generalized anxiety disorder.
To examine the difference between Sana+TAU and TAU on depression symptoms as measured by the Patient Health Questionnaire 9 (PHQ-9) after 28 days. | Baseline, Days 14 and 28
  A self-reported questionnaire for screening and measuring severity of generalized anxiety disorder.
To examine the difference between Sana+TAU compared to TAU on perceived change in quality of life over TAU as measured by the Patient Global Impression of Change scale (PGIC) after 28 days. | Baseline, Days 14 and 28
  A validated tool for screening, diagnosing, monitoring and measuring depression severity and scores each of the 9 Diagnostic and Statistical Manual of Mental Disorder, Fourth Edition (DSM-IV) related criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Acierno, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center
Locations (1):
- Ralph H. Johnson Veteran Affairs Medical Center/Lowcountry Center for Veterans Research, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No